CLINICAL TRIAL: NCT07033182
Title: An Open-Label, Parallel, Single-Dose Study to Assess the Pharmacokinetics and Safety of Levornidazole Disodium Phosphate for Injection in Subjects With Varying Degrees of Renal Impairment
Brief Title: Pharmacokinetics and Safety Study of Levornidazole Disodium Phosphate for Injection in Subjects With Renal Impairment and Normal Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yangtze River Pharmaceutical Group Jiangsu Zilong Pharmaceutical Co. Ltd (Industry)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); Beijing Haisha Consulting Co., Ltd (Unknown)
Responsible Party: Sponsor
Organization: Yangtze River Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YZJ-ZAXZ-403
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Infections Caused by Anaerobic Bacteria; Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group A (Experimental): Severe renal impairment
  Interventions: Drug: Levornidazole Disodium Phosphate for Injection
- Experimental Group B (Experimental): Moderate renal impairment
  Interventions: Drug: Levornidazole Disodium Phosphate for Injection
- Experimental Group C (Experimental): Normal renal function
  Interventions: Drug: Levornidazole Disodium Phosphate for Injection

INTERVENTIONS:
Drug: Levornidazole Disodium Phosphate for Injection — Single dose, IV

SUMMARY:
To evaluate the pharmacokinetics and safety of a single intravenous dose of levornidazole disodium phosphate for injection in subjects with moderate and severe renal impairment and healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

-

Inclusion criteria（Group A and B-Severe Renal Impairment Group and Moderate Renal Impairment Group）:

1. Subjects who are able to understand and willing to complete the study in strict compliance with the clinical protocol and sign the informed consent form.
2. Male or female subjects aged 18-75 years (inclusive).
3. Weight ≥ 50.0 kg for males, or ≥ 45.0 kg for females, and body mass index (BMI) in the range of 19.0 ~ 30.0 kg/m2 (inclusive).
4. Subjects with diagnosis of chronic kidney disease and/or absolute eGFR did not change significantly within 1 month before screening, absolute eGFR met the renal function classification criteria in the corresponding group at screening, severe renal insufficiency, absolute eGFR: 15 ~ 29 mL/min; moderate renal insufficiency, absolute eGFR: 30 ~ 59 mL/min.
5. Subjects of childbearing potential (including partners), voluntarily take appropriate contraceptive measures from 2 weeks before screening to 3 months after dosing.

Inclusion criteria（Group C-Healthy Subject Group）:

1. Subjects who are able to understand and willing to complete the study in strict compliance with the clinical protocol and sign the informed consent form.
2. Male and female subjects aged 18 - 75 years (inclusive) were matched with subjects in groups A and B for age (mean ± 10 years) and gender (mean ± 1 case of gender in groups A and B).
3. Weight ≥ 50.0 kg for males, or ≥ 45.0 kg for females, and body mass index (BMI) in the range of 19.0 ~ 30.0 kg/m2, matched with BMI of subjects in groups A and B(mean ± 15%).
4. Normal renal function, 90 mL/min ≤ absolute eGFR < 130 mL/min.
5. Screening physical examination, vital signs, 12-lead electrocardiogram, laboratory tests, imaging and abdominal ultrasonography results were normal or abnormal but the investigator judged no clinical significance.
6. Subjects of childbearing potential (including partners), voluntarily take appropriate contraceptive measures from 2 weeks before screening to 3 months after dosing.

Exclusion Criteria:

-

Exclusion criteria(Group A and B-Severe Renal Impairment Group and Moderate Renal Impairment Group):

1. Subjects who are known to be allergic to levornidazole phosphate disodium, levornidazole, ornidazole, other nitroimidazoles or their excipients, or have a history of drug or food allergy, or have a history of specific allergic diseases (such as asthma, urticaria, eczema, etc.).
2. Subjects who have special dietary requirements,who cannot accept a unified diet.
3. Subjects who have poor peripheral venous access or cannot tolerate venous puncture or have a history of needle and blood fainting.
4. Subjects who have received renal transplantation and/or require renal dialysis during the study.
5. Subjects combined with cardiovascular, respiratory, digestive, endocrine, malignant tumor, hematopoietic, mental/nervous system serious diseases in addition to the disease causing renal dysfunction itself, which are considered not suitable for participation by the investigator.
6. Subjects with other clinically significant abnormalities except for laboratory tests, physical examination, vital signs, 12-lead electrocardiogram, imaging tests, and abdominal ultrasonography that are judged to be caused by renal insufficiency and its associated diseases, such as ALT (alanine aminotransferase) and/or AST (aspartate aminotransferase) > 2 times the upper limit of normal and/or TBIL (total bilirubin) > 1.5 times the upper limit of normal; Hb (hemoglobin) < 80 g/L; QTc > 450 ms in men and QTc > 470 ms in women.
7. Subjects with poorly controlled hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg) or heart rate > 120 bmp.
8. Patients with diabetic nephropathy HbAlc (glycosylated hemoglobin) > 8.5% or fasting blood glucose > 8.5 mmol/L, or stable treatment regimen for less than 1 month before screening.
9. Subjects with clinically significant abnormalities in any of hepatitis B virus surface antigen, Treponema pallidum-specific antibody, human immunodeficiency virus antibody, hepatitis C virus antibody.
10. Subjects with a history of drug abuse, drug use within 6 months before screening, or positive drug abuse screening.
11. Subjects who frequently consume alcohol within 3 months prior to screening, i.e., consuming more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of 40% spirits, or 150 mL of wine), or who cannot stop using any alcohol products during the study, or alcohol breath test result > 0.0 mg/100 mL.
12. Subjects who have donated blood or experienced massive blood loss (> 400 mL) within 3 months prior to screening, received blood transfusions or used blood products, planned to donate blood during the trial period or within 1 month after the end of the trial.
13. Subjects who have consumed excessive tea, coffee and/or caffeine-containing beverages (more than 8 cups, 1 cup ≈ 250 mL) daily during the 3 months before screening.
14. Subjects smoke an average of 5 or more cigarettes per day within 3 months prior to screening, or those who cannot stop using any tobacco products during the study.
15. Subjects who have participated in any clinical trial within 3 months prior to screening, or plan to participate in other clinical trials during the study.
16. Subjects who have received any surgery or severe trauma that may affect the safety of the trial or the process of drug in vivo within 30 days before screening, or plan to undergo surgery during the study.
17. Subjects who have received vaccination within 30 days prior to screening, or plan to receive vaccination during the study.
18. Subjects who have used any drugs that inhibit or induce hepatic metabolism of drugs within 30 days before administration.
19. Subjects who have used any prescription drugs, over-the-counter drugs, vitamin products, health products or Chinese herbal medicines other than those for the treatment of renal insufficiency and or its concomitant chronic diseases within 14 days before administration.
20. Subjects who started taking new drugs, dosage forms or adjusted current doses for the treatment of chronic kidney disease and its combined chronic diseases within 14 days before administration.
21. Subjects who have consumed grapefruit, pomelo, pitaya, mango and other fruits or related products affecting metabolic enzymes within 7 days before administration.
22. Subjects who have consumed xanthine-rich, caffeine-containing or alcohol-containing beverages or foods (such as animal viscera, coffee, strong tea, chocolate, cola, etc.) within 48 hours before administration.
23. Lactating women, or women who test positive for pregnancy.
24. Subjects with acute illness from screening to prior to administration.
25. Those who, in the opinion of the investigator, are not suitable for inclusion.

Exclusion criteria（Group C-Healthy Subject Group）:

1. Subjects who are known to be allergic to levornidazole phosphate disodium, levornidazole, ornidazole, other nitroimidazoles or their excipients, or have a history of drug or food allergy, or have a history of specific allergic diseases (such as asthma, urticaria, eczema, etc.).
2. Subjects who have special dietary requirements,who cannot accept a unified diet.
3. Subjects who have poor peripheral venous access or cannot tolerate venous puncture or have a history of needle and blood fainting.
4. Subjects who have a history of serious diseases and chronic diseases such as respiratory system, circulatory system, digestive system, urinary system, blood system, endocrine system, immune system, nervous system, mental system.
5. Those who are positive in any index screening of hepatitis B virus surface antigen, Treponema pallidum-specific antibody, human immunodeficiency virus antibody,or hepatitis C virus antibody；
6. Subjects with a history of drug abuse, drug use within 6 months before screening, or positive drug abuse screening;
7. Subjects who frequently consume alcohol within 3 months prior to screening, i.e., consuming more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of 40% spirits, alcohol or 150 mL of wine), or who cannot stop using any alcohol products during the study, or whose alcohol breath test result > 0.0 mg/100 mL;
8. Subjects who have donated blood or experienced massive blood loss (> 400 mL) within 3 months prior to screening, received blood transfusions or used blood products, planned to donate blood during the trial period or within 1 month after the end of the trial;
9. Subjects who have consumed excessive tea, coffee and/or caffeine-containing beverages (more than 8 cups, 1 cup ≈ 250 mL) daily during the 3 months before screening;
10. Subjects smoke an average of 5 or more cigarettes per day within 3 months prior to screening, or those who cannot stop using any tobacco products during the study.
11. Subjects who have participated in any clinical trial within 3 months prior to screening, or plan to participate in other clinical trials during the study.
12. Subjects who have received any surgery or severe trauma that may affect the safety of the trial or the process of drug in vivo within 30 days before screening, or plan to undergo surgery during the study.
13. Subjects who have received vaccination within 30 days prior to screening, or plan to receive vaccination during the study.
14. Subjects who have used any drugs that inhibit or induce hepatic metabolism of drugs within 30 days before administration.
15. Subjects who have taken any prescription drugs, over-the-counter drugs, health products, vitamins, and Chinese herbal medicines within 14 days before administration.
16. Subjects who have consumed grapefruit, pomelo, pitaya, mango and other fruits or related products affecting metabolic enzymes within 7 days before administration.
17. Subjects who have consumed xanthine-rich, caffeine-containing or alcohol-containing beverages or foods (such as animal viscera, coffee, strong tea, chocolate, cola, etc.) within 48 hours before administration.
18. Lactating women, or women who test positive for pregnancy.
19. Subjects with acute illness from screening to prior to administration.
20. Those who, in the opinion of the investigator, are not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-04-07 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-time Curve From Time 0 to the Last Measurable Concentration (AUC0-t) of levornidazole | From Day 1 to Day 5
Area Under the Plasma Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-∞) of levornidazole | From Day 1 to Day 5
Maximum Observed Plasma Concentration (Cmax) of levornidazole | From Day 1 to Day 5
Clearance (CL) of levornidazole | From Day 1 to Day 5
The Volume of Distribution (Vd) of levornidazole | From Day 1 to Day 5
Time of Maximum Observed Plasma Concentration (Tmax) of levornidazole | From Day 1 to Day 5
Apparent Terminal Elimination Half-life (t1/2) of levornidazole | From Day 1 to Day 5
Mean Residence Time (MRT0-t) of levornidazole | From Day 1 to Day 5
Renal Excretion (Ae) of levornidazole | From Day 1 to Day 5
renal clearance (CLR) of levornidazole | From Day 1 to Day 5
Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 to Day 9

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, China